CLINICAL TRIAL: NCT02848274
Title: Prospective Multicenter International Observational Study for Determination of a Cutaneous Lymphoma International Prognostic Index Model and Impact of Major Therapies in Patients With Advanced Mycosis Fungoides and Sézary Syndrome
Brief Title: ID Of Prognostic Factors In Mycosis Fungoides/Sezary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-32652; LYMNHL0134 (Other: OnCore); NCI-2020-00940 (Registry Identifier: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Mycosis Fungoides; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to develop a prognostic index model for the rare disease of mycosis fungoides and sezary syndrome. This will be done by collecting standardized clinical data at various institutions. The investigators hope this will enable the identification of low- and high-risk groups for survival in order to improve patient care and outcome.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of advanced stage MF or SS (Stages IIB - IVB) within 6 months of presentation to the participating center
* Patients that are expected to have care administered at the participating center or jointly with referring physician(s) where follow-up data would be available

Exclusion Criteria

* Patients diagnosed with early stage MF/SS (Stages IA-IIA) before progressing to advanced stage
* Patients diagnosed with advanced MF/SS more than 6 months prior to initial presentation to the participating center
* Exclude one-time consultation type of new patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with advanced stage mycosis fungoides and/or sezary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | date of diagnosis to death from any cause, up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Kim, MD, Principal Investigator — Stanford University
Locations (13):
- United States (7):
  - City of Hope, Duarte, California
  - Stanford University, School of Medicine, Palo Alto, California
  - University of Iowa, Iowa City, Iowa
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Peter MacCallum Cancer Center,, Melbourne, Australia
- University of Sao Paulo Medical School, São Paulo, Brazil
- Peking University First Hospital, Beijing, China
- The University of Tokyo, Tokyo, Japan
- University Hospitals Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Scarisbrick JJ, Quaglino P, Whittaker S, Bagot M, Guenova E, Papadavid E, Prince HM, Sanches JA, Miyashiro DR, Servitje O, Querfeld C, Akilov O, Arumainathan A, Bennett L, Battistella M, Benstead K, Berti E, Beylot-Barry M, Busschots AM, Cowan R, Dummer R, Dunnill G, Estrach T, Evison F, Bashir A, Geskin L, Gru A, Guitart J, Herrera MC, Hodak E, Horwitz S, Jonak C, Klemke CD, Knobler R, Mckay P, Marschalko M, Massone C, Matin R, Mitteldorf C, Novoa R, Ortiz-Romero P, Pimpinelli N, Pujol RM, Ranki A, Vakeva L, Rieger KE, Stadler R, Trautinger F, Latzka J, Vermeer M, Wachsmuth R, Weatherhead S, Wehkamp U, Wobser M, Kim YH. A new prognostic index (CLIPI) for advanced cutaneous lymphoma enables precise patient risk stratification. Blood. 2025 Oct 2;146(14):1687-1692. doi: 10.1182/blood.2025029628. PMID 40663780